CLINICAL TRIAL: NCT05982886
Title: Biomarker Testing and Treatment Patterns Among Patients With PIK3CA Mutation in Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719A0US11
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer,; PIK3CA,; Alpelisib,; non-interventional study,; HR+
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- PIK3CA positive: HR+ Her2-
- PIK3CA positive: HR- Her2-
- PIK3CA positive: HR- Her2+
- PIK3CA positive: HR+ Her2+
- PIK3CA negative

SUMMARY:
This was a retrospective observational study of patients with advanced breast cancer (BC). This non-interventional study was conducted using discrete structured data and medical record abstraction, if needed, from patients treated at Texas Oncology, the designated research organization and a community oncology practice. The first date of a new diagnosis of advanced BC (de novo or progressed to advanced BC) defined the study index date. To allow for an adequate potential duration of follow-up (retrospectively observed) after the index date over which PIK3CA testing and treatment patterns was observed, a minimum follow-up opportunity of 6 months after the diagnosis of advanced BC at the time of data pull and/or abstraction was required.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the following criteria were eligible for abstraction:
* Newly diagnosed advanced BC between 01 January 2015, and 30 June 2020
* Evaluated for a PIK3CA mutation and identified PIK3CA gene status
* No evidence of active other malignant neoplasms within 3 years (except nonmelanoma skin cancer or carcinoma in situ) prior to diagnosis of advanced BC
* At least 18 years of age at the time of first diagnosis of BC
* Patients may be alive or deceased at the time of abstraction
* Not ever enrolled in the following interventional clinical trials evaluating PI3K inhibitors:

  * SOLAR-1 trial (NCT0243731) evaluating alpelisib (BYL719)
  * BELLE-2 or BELLE-3 trial (NCT01610284, NCT01633060) evaluating buparlisib (BKM120)
  * SANDPIPER trial (NCT02340221) evaluating taselisib (GDC-0032)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 1093 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with PIK3CA mutations | Up to approximately 6 years
Time from first BC diagnosis to first PIK3CA evaluation | Up to approximately 6 years
Time from advanced BC diagnosis to first PIK3CA evaluation | Up to approximately 6 years
Time from initiation of first-line treatment for advanced BC diagnosis to first PIK3CA evaluation | Up to approximately 6 years
Number of tests for patients with CDK4/6 inhibitor treatment | Up to approximately 6 years
Time from progression on CDK4/6 inhibitor to first PIK3CA evaluation | Up to approximately 6 years
Year of (first, where applicable) PIK3CA evaluation | Up to approximately 6 years
Result of PIK3CA evaluation (negative, positive, unknown) | Up to approximately 6 years
Type of biopsy | Up to approximately 6 years
Type of tissue sample, for patients who had tissue biopsy | Up to approximately 6 years
Source of tissue sample, for patients who had tissue biopsy | Up to approximately 6 years
Analytical method used for PIK3CA evaluation | Up to approximately 6 years

SECONDARY OUTCOMES:
Age at advanced breast cancer diagnosis | Up to approximately 6 years
Stage when patients were diagnosed with BC | Up to approximately 6 years
Number of patients with known metastatic sites | Up to approximately 6 years
Performance as assessed by Karnofsky Performace Scale | Up to approximately 6 years
  The Karnofsky Performance Scale is a measure of functional impairment.
Performance as assessed by the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale | Up to approximately 6 years
  The ECOG performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
Height | Up to approximately 6 years
Weight | Up to approximately 6 years
Body mass index (BMI) | Up to approximately 6 years
Number of patients per stage of cancer | Up to approximately 6 years
Number of patients per line of treatment | Up to approximately 6 years
Time from advanced diagnosis to initiation of lines of treatment | Up to approximately 6 years
Number of patients per systemic therapy | Up to approximately 6 years
Number of patients per treatment sequence | Up to approximately 6 years
Number of patients per supportive treatment | Up to approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States